CLINICAL TRIAL: NCT06831188
Title: The Effect Of Exercise On Performance And Quality Of Life In Children With Autism Spectrum Disorder
Brief Title: Exercise Efficacy on Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Şensu Dinçer, Medical doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: autism spectrum disorder-SY
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: autism; exercise; MOBAK-1; 6-min walk test
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- specific type exercise group (Experimental): The participants will be given exercise programs for 12 weeks, and these exercises will be performed regularly.
  Interventions: Other: specific type exercise group
- daily life exercise group (Active Comparator): - random games which includes physical activity
  Interventions: Other: daily life exercise group

INTERVENTIONS:
Other: daily life exercise group — random games which includes physical activity
  Arms: daily life exercise group
Other: specific type exercise group — 10 minutesTreadmill Walk, Playdough or ball squeeze, Towel wring,Throwing to target, catching the tennis ball, bouncing a ball inside borders without losing control, dribbling a ball inside borders without losing control, tandem walk, Single leg stance balance on balance pad or pillow, rolling forward, Jumping exercises, Side stepping, etc
  Arms: specific type exercise group

SUMMARY:
The goal of this clinical trial is to learn if regular exercise intervention may improve the health status of the participants diagnosed with autism spectrum disorder, ages between 5-13 years old. The main question it aims to answer is:

* if combined regular exercise program improves motor skills, repetitive movements, aerobic capacity and quality of life of participants?
* Researchers will compare the exercising and non-exercising participants to see if regular exercise improves the health related parameters.

Participants will do exercise for 12 weeks regularly.

DETAILED DESCRIPTION:
Before and after the exercise program;

* the parents of the participants will fill out the ABC problem behaviour control scale
* the participants will perform 6 minute walk test, sit-reach flexibility test, grip strength test. Body fat analysis will be performed by using Bioimpedance Analysis Method.
* participants will also perform MoBAK-1 test which measures motor competencies

Exercise program include; 10 minutesTreadmill Walk, Playdough or ball squeeze, Towel wring,Throwing to target, catching the tennis ball, bouncing a ball inside borders without losing control, dribbling a ball inside borders without losing control, tandem walk, Single leg stance balance on balance pad or pillow, rolling forward, Jumping exercises, Side stepping, etc.

The implementation of exercise programs, the follow-up process, and data recording methods will be documented and applied by the research team.

Data will be analyzed in the SPSS 28 statistical package program. The data distribution will be checked by Kolmogorov Smirnov and the homogeneity of variances by the Levene test. For variables with normal distribution, One-Way ANOVA will be used for multiple comparisons, and an Independent t-test will be used for pairwise comparisons. Wilcoxon test will be used for pairwise comparisons in dependent variables that do not fit a normal distribution, and the Mann- Whitney U test will be used in independent variables. The relationship between continuous variables will be tested using the correlation coefficient, and the relationship between categorical variables will be tested using the chi-square test. Descriptive statistics will be given as mean ± standard deviation. Results will be considered statistically significant for p<0.05.

ELIGIBILITY:
Inclusion Criteria: children with autism spectrum disorder

-

Exclusion Criteria:

* children who are unable to adapt exercise programs

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | Through study completion, an average of 12 weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance.
sit-reach test reach flexibility test | Through study completion, an average of 12 weeks
  The Sit and reach test is one of the linear flexibility tests which helps to measure the extensibility of the hamstrings and lower back
grip strength | Through study completion, an average of 12 weeks
  Grip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It can be used as a screening tool for the measurement of upper body strength and overall strength.
body composition analyses | Through study completion, an average of 12 weeks
  Body fat percentage will be measured by using Bioimpedance measurement system
MOBAK-1 basic motor competencies | Through study completion, an average of 12 weeks
  The MOBAK 1 test battery is a recent instrument developed to assess motor competence in primary physical education.The MOBAK-1 testing battery has been r developed with the aim of assessing a wide panel of motor skills in relationship with body movement and object-control abilities

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)